CLINICAL TRIAL: NCT05150912
Title: Manual Therapy Based on Neurodynamic Techniques Versus Manual Therapy Including Desensitization Maneuvers With One Year Follow-up :Randomized Clinical Trial
Brief Title: Mnaual Therapy in Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sahar Ahmed Abdalbary, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nahda University
Record Dates: First submitted 2021-11-15; First posted 2021-12-09 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuro dynamic (Active Comparator): Neurodynamic techniques.
  Interventions: Other: Manual therapy
- desensitization (Active Comparator): Desensitization maneuvers
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — strching neck

SUMMARY:
2 groups of patients randomized for the treatment.

DETAILED DESCRIPTION:
One group treated with neurodynamic techniques and the the other with the desensitization maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Pain and paresthesia at median nerve distribution ,positive tinel sign and positive phalen sign.

Exclusion Criteria:

* Any sensory and/or motor deficit in either ulnar or radial nerve
* age greater than 55 years .
* male sex.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 412 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
PAIN and function | after one year
  Boston carpal tunnel questionnaire (BCTQ) measure function and pain
muscle strength | 3 month
  measured by dynamometer to measure cylindrical grip and pincer grip

CONTACTS AND LOCATIONS:
Locations (1):
- Sahar, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No